CLINICAL TRIAL: NCT03086343
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Study Comparing Upadacitinib (ABT-494) to Abatacept in Subjects With Moderately to Severely Active Rheumatoid Arthritis With Inadequate Response or Intolerance to Biologic DMARDs (bDMARDs) on Stable Conventional Synthetic Disease Modifying Anti-Rheumatic Drugs (csDMARDs)
Brief Title: A Phase 3 Study to Compare Upadacitinib to Abatacept in Subjects With Rheumatoid Arthritis on Stable Dose of Conventional Synthetic Disease- Modifying Antirheumatic Drugs (csDMARDs) Who Have an Inadequate Response or Intolerance to Biologic DMARDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-925; 2016-000933-37 (EudraCT Number)
Record Dates: First submitted 2017-03-20; First posted 2017-03-22 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Musculoskeletal Disease; Arthritis; Joint Disease; Anti-inflammatory agents; Antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — Abatacept; Sodium Chloride; Solutions; upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Primary Cohort: Abatacept/Upadacitinib 15 mg QD (Active Comparator): Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20. Period 2: open label upadacitinib 15 mg QD for 192 weeks.
  Interventions: Drug: Abatacept; Drug: Upadacitinib; Drug: Placebo for upadacitinib
- Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD (Experimental): Period 1: One 15 mg upadacitinib oral tablet QD for 24 weeks. Period 2: open label upadacitinib 15 mg QD for 192 weeks.
  Interventions: Drug: Placebo for abatacept (0.9% Sodium Chloride Injection or Solution for Infusion); Drug: Upadacitinib
- 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD (Experimental): Period 1: One upadacitinib 30 mg oral tablet QD for 24 weeks. Period 2: open label upadacitinib 30 mg (reduced to 15 mg per Amendment 5) QD for 192 weeks.
  Interventions: Drug: Placebo for abatacept (0.9% Sodium Chloride Injection or Solution for Infusion); Drug: Upadacitinib
- 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD (Active Comparator): Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20. Period 2: open label upadacitinib 30 mg (reduced to 15 mg per Amendment 5) QD for 192 weeks.
  Interventions: Drug: Abatacept; Drug: Upadacitinib; Drug: Placebo for upadacitinib

INTERVENTIONS:
Drug: Abatacept — IV infusion
  Arms: 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD; Primary Cohort: Abatacept/Upadacitinib 15 mg QD
Drug: Placebo for abatacept (0.9% Sodium Chloride Injection or Solution for Infusion) — IV infusion
  Arms: 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD; Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD
Drug: Upadacitinib — 15 mg extended release tablet
  Other Names: ABT-494
Drug: Placebo for upadacitinib — Film-coated tablet
  Arms: 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD; Primary Cohort: Abatacept/Upadacitinib 15 mg QD

SUMMARY:
The study objective of Period 1 was to compare the safety and efficacy of upadacitinib 15 mg once daily (QD) to abatacept on a background of conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) for the treatment of signs and symptoms of rheumatoid arthritis (RA) in biologic disease-modifying antirheumatic drug (bDMARD)-inadequate response or bDMARD-intolerant participants with moderately to severely active RA. The study objective of Period 2 is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 15 mg QD in participants with RA who had completed Period 1.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter study with 2 periods. Period 1 was a 24-week, randomized, double-blind, parallel-group, active-controlled period designed to compare the safety and efficacy of upadacitinib 15 mg and abatacept for the treatment of signs and symptoms of participants with moderately to severely active RA who had an inadequate response to or intolerance to bDMARD therapy and were currently on a stable dose of csDMARD(s) and had never received abatacept. Period 2 is an open-label, long-term extension study to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 15 mg once a day (QD) in participants with RA who had completed Period 1.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for ≥ 3 months who also fulfill the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA
* Participants have been treated for ≥ 3 months prior to the screening visit with ≥ 1 bDMARD therapy, but continue to exhibit active RA or had to discontinue due to intolerability or toxicity, irrespective of treatment duration and have never received abatacept prior to the first dose of study drug
* Participants have been receiving csDMARD therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug. The following csDMARDs are allowed: methotrexate (MTX), sulfasalazine, hydroxychloroquine, chloroquine, and leflunomide. A combination of up to two background csDMARDs is allowed except the combination of MTX and leflunomide
* Meets the following criteria: ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits and high-sensitivity C-reactive protein (hsCRP) ≥ 3 mg/L at Screening

Main Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to upadacitinib, tofacitinib, baricitinib and filgotinib)
* Prior exposure to abatacept
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA. Current diagnosis of secondary Sjogren's Syndrome is permitted
* Laboratory values meeting the following criteria within the Screening period prior to the first dose of study drug: serum aspartate transaminase > 2 × upper limit of normal (ULN); serum alanine transaminase > 2 × ULN; estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease formula < 40 mL/minute/1.73 meter (m)^2; total white blood cell count < 2,500/ μL; absolute neutrophil count < 1,500/μL; platelet count < 100,000/μL; absolute lymphocyte count < 800/μL; and hemoglobin < 10 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (161):
- United States (44):
  - SunValley Arthritis Center, Lt /ID# 154558, Peoria, Arizona
  - AZ Arthritis & Rheum Research /ID# 156539, Sun City, Arizona
  - AZ Arth & Rheum Res /ID# 167161, Tucson, Arizona
  - CHI St. Vincent Medical Group /ID# 154561, Hot Springs, Arkansas
  - Saint Jude Heritage /ID# 158833, Fullerton, California
  - Kotha and Kotha /ID# 154573, La Mesa, California
  - Denver Arthritis Clinic /ID# 159195, Denver, Colorado
  - Arthritis and Rheum Clin N. CO /ID# 155673, Fort Collins, Colorado
  - Scientia Medical Research /ID# 159189, Lakewood, Colorado
  - Clinical Res of West FL, Inc. /ID# 154576, Clearwater, Florida
  - Advanced Clin Res of Orlando /ID# 154580, Ocoee, Florida
  - Gulf Region Clinical Res Inst /ID# 154597, Pensacola, Florida
  - W. Broward Rheum Assoc Inc. /ID# 158835, Tamarac, Florida
  - Lovelace Scientific Resources /ID# 154600, Venice, Florida
  - Jefrey D. Lieberman, MD, P.C. /ID# 157178, Decatur, Georgia
  - Advanced Clinical Research /ID# 154603, Meridian, Idaho
  - PMG Research of Christie Clini /ID# 154569, Champaign, Illinois
  - Bluegrass Community Research /ID# 154604, Lexington, Kentucky
  - Four Rivers Clinical Research /ID# 154606, Paducah, Kentucky
  - Ochsner Clinic Foundation /ID# 154585, Baton Rouge, Louisiana
  - The Center for Rheumatology & Bone Research /ID# 158723, Wheaton, Maryland
  - West Michigan Rheumatology /ID# 154551, Grand Rapids, Michigan
  - Advanced Rheumatology, PC /ID# 154589, Lansing, Michigan
  - Clinvest Research LLC /ID# 154554, Springfield, Missouri
  - Overlook Medical Center /ID# 154794, Summit, New Jersey
  - Atlantic Coast Research /ID# 155234, Toms River, New Jersey
  - Ocean Rheumatology, PA /ID# 162980, Toms River, New Jersey
  - Arthritis and Osteo Assoc /ID# 154560, Las Cruces, New Mexico
  - The Center for Rheumatology /ID# 162979, Albany, New York
  - NYU Langone Rheum Assoc /ID# 155236, Lake Success, New York
  - NYU Langone Medical Center /ID# 158829, New York, New York
  - Physicians East, PA /ID# 154565, Greenville, North Carolina
  - PMG Research of Salisbury /ID# 154605, Salisbury, North Carolina
  - PMG Research of Wilmington LLC /ID# 154584, Wilmington, North Carolina
  - Wake Forest Baptist Medical Center /ID# 154586, Winston-Salem, North Carolina
  - Oregon Health and Science University /ID# 163822, Portland, Oregon
  - East Penn Rheumatology Assoc /ID# 159193, Bethlehem, Pennsylvania
  - Altoona Ctr Clinical Res /ID# 154572, Duncansville, Pennsylvania
  - University of Pittsburgh MC /ID# 157434, Pittsburgh, Pennsylvania
  - West Tennessee Research Inst /ID# 158721, Jackson, Tennessee
  - Adriana Pop-Moody MD Clinic PA /ID# 154607, Corpus Christi, Texas
  - P&I Clinical Research /ID# 159191, Lufkin, Texas
  - DM Clinical Research /ID# 158722, Tomball, Texas
  - Care Access Research /ID# 158098, Salt Lake City, Utah
- Argentina (9):
  - Aprillus Asistencia e Investig /ID# 159173, Capital Federal, Buenos Aires
  - Ctr Privado Med Familiar /ID# 158814, Buenos Aires
  - Atencion Integral en Reuma /ID# 155696, Buenos Aires
  - Hospital General de Agudos /ID# 167117, Buenos Aires
  - Inst. de Rehab. Psicofisica /ID# 167768, CABA
  - Inst. Rheumatologic Strusberg /ID# 159021, Córdoba
  - Instituto Medico DAMIC /ID# 167770, Córdoba
  - DIM Clinica Privada /ID# 167769, Ramos Mejía
  - Instituto CAICI SRL /ID# 159022, Rosario, Santa FE
- Australia (3):
  - Rheumatology Research Unit /ID# 159174, Maroochydore, Queensland
  - The Queen Elizabeth Hospital /ID# 159175, Woodville, South Australia
  - Western Health Footscray Hospi /ID# 157968, Footscray, Victoria
- CHU UCL Namur /ID# 157628, Namur, Belgium
- Brazil (8):
  - CEDOES-Centro de Diagnóstico e Pesquisa da Osteoporose do Espírito Santo LTDA /ID# 155228, Vitória, Espírito Santo
  - Santa Casa de Belo Horizonte /ID# 154631, Belo Horizonte, Minas Gerais
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 154564, Juiz de Fora, Minas Gerais
  - Ceti - Centro de Estudos Em Terapias Inovadoras Ltda /Id# 154634, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 161211, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 159176, Porto Alegre, Rio Grande do Sul
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos /ID# 154632, Santo André, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda /ID# 159587, São Paulo, São Paulo
- Bulgaria (4):
  - MHAT Trimontsium /ID# 155226, Plovdiv
  - Diag Consult Ctr 17 Sofia EOOD /ID# 169298, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 155000, Sofia
  - Medical Centre Synexus Sofia /ID# 201807, Sofia
- Canada (4):
  - The Waterside Clinic /ID# 159178, Barrie, Ontario
  - Adachi Medicine Prof. Corp /ID# 158024, Hamilton, Ontario
  - Institut de Rhum. de Montreal /ID# 155001, Montreal, Quebec
  - Groupe de Recherche en Maladies Osseuses /ID# 154601, Sainte-Foy, Quebec
- Czechia (2):
  - Revmatologicky ustav Praha /ID# 154612, Prague, Praha 2
  - Medical Plus, s.r.o. /ID# 155230, Uherské Hradište
- Germany (4):
  - Uniklinik Koln /ID# 156047, Cologne, North Rhine-Westphalia
  - Praxis fuer Rheumatologie /ID# 156156, Berlin
  - Rheumaforschungszentrum II /ID# 157177, Hamburg
  - Welcker, Planegg, DE /ID# 160185, Planegg
- University General Hospital of Heraklion "PA.G.N.I" /ID# 163916, Heraklion, Greece
- Hungary (5):
  - Budai Irgalmasrendi Korhaz /ID# 154457, Budapest
  - Obudai Egeszsegugyi Centrum Kft. /ID# 156159, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 159183, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet /ID# 159689, Eger
  - MAV Korhaz ess Rendelointezet /ID# 154455, Szolnok
- Our Lady's Hospital /ID# 161149, Manorhamilton, Ireland
- Israel (4):
  - Barzilai Medical Center /ID# 161685, Ashkelon
  - The Lady Davis Carmel MC /ID# 161686, Haifa
  - Meir Medical Center /ID# 162774, Kfar Saba
  - Sheba Medical Center /ID# 163154, Ramat Gan
- Italy (6):
  - Istituto Clinico Humanitas /ID# 154999, Rozzano, Milano
  - AOU Citta della Salute Scienza /ID# 154577, Turin, Piedmont
  - Presidio Columbus, Fondazione Policlinico Gemelli Universita Cattolica S. Cuore /ID# 162252, Rome, Roma
  - A.O. Univ. Ospedali Riuniti /ID# 161707, Ancona, The Marches
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele /ID# 161172, Catania
  - ASST G. Pini /ID# 162223, Milan
- Latvia (2):
  - D.Saulites-Kandevicas PP /ID# 154578, Liepāja
  - Riga East Clinical Univ Hosp /ID# 155024, Riga
- Mexico (5):
  - Morales Vargas Centro de Investigacion S.C. /ID# 200800, León, Guanajuato
  - Centro Integral en Reumatología S.A de C.V /ID# 204493, Guadalajara, Jalisco
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 154579, Mexico City, Mexico City
  - RM Pharma Specialists S.A de C.V /ID# 159588, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevención de Enfermedades Cardiova /ID# 160126, Mexico City
- Netherlands (4):
  - Antonius Ziekenhuis /ID# 155737, Sneek, Provincie Friesland
  - Reade /ID# 161002, Amsterdam
  - Spaarne Gasthuis /ID# 161003, Haarlem
  - Medisch Centrum Leeuwarden /ID# 156043, Leeuwarden
- New Zealand (2):
  - Timaru Medical Specialists Ltd /ID# 159184, Timaru
  - Wellington Hospital (Capital and Coast District Health Board) /ID# 154591, Wellington
- Poland (8):
  - Medyczne Centrum Hetmanska /ID# 155746, Poznan, Greater Poland Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 157180, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne AMED Warszawa Targowek /ID# 159589, Warsaw, Masovian Voivodeship
  - Gabinet Internistyczno Reum. /ID# 157433, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j. /ID# 202998, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni /ID# 202472, Gdynia, Pomeranian Voivodeship
  - Centrum Med Amed Oddzial Lodzi /ID# 154458, Lodz
  - Salve Medica Sp. z o.o. S.K. /ID# 202473, Lodz, Łódź Voivodeship
- Portugal (6):
  - Instituto Portugues De Reumatologia /ID# 155698, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 200035, Lisbon, Lisbon District
  - Hospital Garcia de Orta, E.P.E /ID# 164056, Almada, Setúbal District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 200037, Lisbon
  - Unidade Local De Saude Do Alto Minho /ID# 200036, Viana do Castelo
  - Centro Hosp de Tondela-Viseu /ID# 155699, Viseu
- Puerto Rico (2):
  - Dr. Ramon L. Ortega-Colon, MD /ID# 158097, Carolina
  - GCM Medical Group /ID# 156158, San Juan
- Romania (2):
  - Spitalul Clinic Dr. I. Cantacuzino /ID# 155893, Bucharest, București
  - Spitalul Clinic Sf. Maria /ID# 167245, Bucharest
- Russia (5):
  - Family Outpatient clinic#4 LLC /ID# 203524, Korolev, Moscow
  - LLC Medical Center /ID# 203523, Novosibirsk, Novosibirsk Oblast
  - Alliance Biomedical Ural Group /ID# 154609, Izhevsk, Udmurtiya Republic
  - State Budget Healthcare Instit /ID# 154593, Moscow
  - Nort-Western State Medical Uni /ID# 154610, Saint Petersburg
- Slovakia (3):
  - Novamed,spol.s.r.o. /ID# 157928, Banská Bystrica
  - Univerzitna Nemocnica Bratislava /ID# 161143, Bratislava
  - Narodny ustav reumatickych chorob Piestany /ID# 156864, Pieštany
- South Korea (3):
  - SMG-SNU Boramae Medical Center /ID# 155788, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido St. Mary's Hospital /ID# 155231, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 154639, Seoul
- Spain (6):
  - Hospital Universitario Reina S /ID# 155701, Córdoba
  - Hospital General Univ de Elche /ID# 158825, Elche
  - Hospital Universitario La Paz /ID# 163636, Madrid
  - Corp Sanitaria Parc Tauli /ID# 163634, Sabadell, Barcelona
  - Complejo Hospitalario /ID# 155700, Santiago de Compostela
  - Hospital Infanta Luisa /ID# 154641, Seville
- Sweden (4):
  - Skanes Universitetssjukhus /ID# 165133, Malmo, Skåne County
  - Akademiskt specialistcentrum Centrum for reumatologi /ID# 156046, Stockholm, Stockholm County
  - Sahlgrenska University Hosp /ID# 162775, Gothenburg
  - Vastmanlands Sjukhus /ID# 159186, Västerås
- Switzerland (4):
  - Hopitaux Universitaires de Geneve /ID# 159083, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen /ID# 155232, Sankt Gallen, Canton of St. Gallen
  - University Hospital of Basel /ID# 160860, Basel
  - HFR Fribourg - Hopital Canton /ID# 160970, Fribourg
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty /ID# 167995, Ankara
  - Ankara Univ Medical Faculty /ID# 162691, Ankara
  - Akdeniz University Faculty /ID# 163153, Antalya
  - Istanbul Fizik Tedavi Rehabilitasyon Egitim ve Arastırma Hastanesi /ID# 169479, Istanbul
- United Kingdom (5):
  - Whipps Cross Univ Hospital /ID# 205985, London, London, City of
  - Ninewells Hospital /ID# 156050, Dundee
  - Altnagelvin Area Hospital /ID# 156540, Londonderry
  - Lancashire Care NHS Foundation /ID# 156042, Preston
  - Royal Cornwall Hospital /ID# 157785, Truro

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Rubbert-Roth A, Enejosa J, Pangan AL, Haraoui B, Rischmueller M, Khan N, Zhang Y, Martin N, Xavier RM. Trial of Upadacitinib or Abatacept in Rheumatoid Arthritis. N Engl J Med. 2020 Oct 15;383(16):1511-1521. doi: 10.1056/NEJMoa2008250. PMID 33053283
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Rubbert-Roth A, Kato K, Haraoui B, Rischmueller M, Liu Y, Khan N, Camp HS, Xavier RM. Safety and Efficacy of Upadacitinib in Patients with Rheumatoid Arthritis Refractory to Biologic DMARDs: Results Through Week 216 from the SELECT-CHOICE Study. Rheumatol Ther. 2024 Oct;11(5):1197-1215. doi: 10.1007/s40744-024-00694-x. Epub 2024 Jul 20. PMID 39031276
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Tundia N, Martin N, Suboticki JL, Patel J, Goldschmidt D, Song Y, Wright GC. Patient-reported outcomes of upadacitinib versus abatacept in patients with rheumatoid arthritis and an inadequate response to biologic disease-modifying antirheumatic drugs: 12- and 24-week results of a phase 3 trial. Arthritis Res Ther. 2022 Jun 24;24(1):155. doi: 10.1186/s13075-022-02813-x. PMID 35751108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had a 24-week, randomized, double-blind, parallel-group, active-controlled period (Period 1) and an open-label long-term extension study (Period 2).
  Primary Cohort: Participants enrolled under Amendment 4 or 3.01, randomized to upadacitinib 15 mg once daily (QD) or abatacept intravenous (IV)/upadacitinib 15 mg QD.
Pre-assignment Details: 30 mg Cohort: Participants enrolled under Amendment 3, randomized to upadacitinib 30 mg QD or abatacept IV/upadacitinib 30 mg QD. Starting with Amendment 5, all participants received open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.
  One participant who was a screen failure was randomized in error and did not receive study drug (and is not included in any data table).
Period: Period 1
Arm/Group | Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD | Primary Cohort: Abatacept/Upadacitinib 15 mg QD | 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD | 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD
Started | 303 | 309 | 21 | 23
Completed | 278 | 277 | 18 | 21
Not Completed | 25 | 32 | 3 | 2
Not completed — Adverse Event | 7 | 7 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 10 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 0
Not completed — Other, Not Specified | 10 | 12 | 2 | 1
Not completed — Missing | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD | Primary Cohort: Abatacept/Upadacitinib 15 mg QD | 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD | 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD
Started | 277 (Includes participants who entered Period 2 study participation without study drug.) | 277 (Includes participants who entered Period 2 study participation without study drug.) | 17 (Includes participants who entered Period 2 study participation without study drug.) | 20 (Includes participants who entered Period 2 study participation without study drug.)
Entered Period 2 on Study Drug | 271 | 276 | 17 | 19
Upadacitinib Dose Switch From 30 mg QD to 15 mg QD During Part 2 | 0 | 0 | 12 | 12
No Upadacitinib Dose Switch During Part 2 | 0 | 0 | 5 | 7
Completed | 207 | 208 | 11 | 12
Not Completed | 70 | 69 | 6 | 8
Not completed — Adverse Event | 20 | 11 | 1 | 2
Not completed — Withdrawal by Subject | 15 | 25 | 2 | 2
Not completed — Lost to Follow-up | 6 | 11 | 1 | 0
Not completed — COVID-19 Infection | 5 | 0 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 1 | 0 | 0 | 0
Not completed — Other, Not Specified | 23 | 22 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least one dose of study drug during Period 1
Groups:
- Primary Cohort: Upadacitinib 15 mg QD: Period 1: One 15 mg upadacitinib oral tablet QD for 24 weeks.
- Primary Cohort: Abatacept; 30 mg Cohort: Abatacept: Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20.
- 30 mg Cohort: Upadacitinib 30 mg QD: Period 1: One upadacitinib 30 mg oral tablet QD for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort: Upadacitinib 15 mg QD | Primary Cohort: Abatacept | 30 mg Cohort: Upadacitinib 30 mg QD | 30 mg Cohort: Abatacept | Total
Number analyzed (Participants) | 303 | 309 | 21 | 23 | 656
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 30 | 31 | 5 | 2 | 68
  40 - 64 years | 209 | 207 | 10 | 17 | 443
  ≥ 65 years | 64 | 71 | 6 | 4 | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 253 | 16 | 20 | 538
  Male | 54 | 56 | 5 | 3 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 112 | 117 | 4 | 5 | 238
  Not Hispanic or Latino | 191 | 192 | 17 | 18 | 418
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 288 | 285 | 19 | 20 | 612
  Black or African American | 7 | 14 | 2 | 3 | 26
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 0 | 0 | 11
  Multiple | 2 | 2 | 0 | 0 | 4
  Other | 0 | 0 | 0 | 0 | 0
Geographic Region [Count of Participants; unit: Participants]
  North America | 72 | 73 | 14 | 16 | 175
  South/Central America | 98 | 99 | 0 | 0 | 197
  Western Europe | 43 | 45 | 1 | 1 | 90
  Eastern Europe | 77 | 77 | 6 | 6 | 166
  Asia | 4 | 4 | 0 | 0 | 8
  Other | 9 | 11 | 0 | 0 | 20
Disease Activity Score Based on C-reactive protein (CRP; DAS28 [CRP]) [Count of Participants; unit: Participants] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission.
  Participants
    Score > 5.1 | 224 | 241 | 15 | 19 | 499
    Score ≤ 5.1 | 79 | 67 | 4 | 3 | 153
    Score Missing | 0 | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score (DAS) 28 C-Reactive Protein (CRP) at Week 12 (Non-inferiority)
Description: The Disease Activity Score (DAS) 28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study drug; multiple imputation was used for missing data. (The Statistical Analysis Plan (SAP) excluded the the 30 mg Cohorts from these efficacy analyses.)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Upadacitinib 15 mg: One 15 mg tablet taken once per day by mouth for 24 weeks
- Abatacept: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) intravenous (IV) infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20
Arm/Group | Upadacitinib 15 mg | Abatacept
Number analyzed (Participants) | 303 | 309
units on a scale | -2.52 [-2.66 to -2.37] | -2.00 [-2.14 to -1.85]
Statistical Analysis 1: Comparison: Upadacitinib 15 mg vs Abatacept; In order to preserve Type I error, a step-down approach was used to test the primary and ranked secondary endpoints in a pre-specified order where statistical significance at the 0.05 level could be claimed for a lower ranked endpoint only if the previous endpoint in the sequence met the requirements of significance; Test type: Non-Inferiority — The non-inferiority of upadacitinib 15 mg versus abatacept was tested using the 95% confidence interval (CI) of treatment difference against a non-inferiority margin of 0.6; p < 0.001, ANCOVA — The ANCOVA model included treatment as the fixed factor; corresponding baseline value and the stratification factor of prior bDMARD used as covariates; LS Mean Difference = -0.52, 95% CI 2-sided [-0.69 to -0.35] — Treatment Difference = Upadacitinib 15 mg - Abatacept

2. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28 C-Reactive Protein (CRP) at Week 12 (Superiority)
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Upadacitinib 15 mg | Abatacept
Number analyzed (Participants) | 303 | 309
units on a scale | -2.52 [-2.66 to -2.37] | -2.00 [-2.14 to -1.85]
Statistical Analysis 1: Comparison: Upadacitinib 15 mg vs Abatacept; In order to preserve Type I error, a step-down approach was used to test the primary and ranked secondary endpoints in a pre specified order where statistical significance at the 0.05 level could be claimed for a lower ranked endpoint only if the previous endpoint in the sequence met the requirements of significance; Test type: Superiority; p < 0.001, ANCOVA — This comparison was a ranked secondary endpoint in the pre-specified multiplicity testing sequence; The ANCOVA model included treatment as the fixed factor; corresponding baseline value and the stratification factor of prior bDMARD used as covariates; LS Mean Difference = -0.52, 95% CI 2-sided [-0.69 to -0.35] — Treatment Difference = Upadacitinib 15 mg - Abatacept

3. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Disease Activity Score (DAS) 28 C-Reactive Protein (CRP) at Week 12 (Superiority)
Description: The Disease Activity Score (DAS) 28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS 28 score less than 2.6 indicates clinical remission.
Time Frame: At Week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study drug; participants who prematurely discontinued study drug were considered non-responders after discontinuation. (The Statistical Analysis Plan (SAP) excluded the the 30 mg Cohorts from these efficacy analyses.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 15 mg | Abatacept
Number analyzed (Participants) | 303 | 309
percentage of participants | 30.0 [24.9 to 35.2] | 13.3 [9.5 to 17.1]
Statistical Analysis 1: Comparison: Upadacitinib 15 mg vs Abatacept; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was a ranked secondary endpoint in the pre-specified multiplicity testing sequence; The stratification factor of prior failed bDMARD was used; Mean Difference = 16.8, 95% CI 2-sided [10.4 to 23.2] — Treatment Difference = Upadacitinib 15 mg - Abatacept

ADVERSE EVENTS:
Time Frame: All Cause Mortality: From informed consent through the end of study. Period 1, all arms: median of 168 days. Period 2, Upa 15 mg only arms: median of 1374 days; Upa 30 mg only arms: median of 925 days; Abatacept/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD arm: median of 450 days; Upadacitinib 30 mg QD/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD arm: median of 446.5 days.
Description: Adverse Event Time Frame: From informed consent until discontinuation of study drug administration (up to 24 weeks for Period 1 and up to 192 weeks for Period 2), plus 70 days.
  Per protocol, for analysis of Period 1 safety data, the Primary and 30 mg Cohorts receiving abatacept were combined.
Groups:
- Period 1, Primary and 30 mg Cohorts: Abatacept: Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20.
- Period 1, Primary Cohort: Upadacitinib 15 mg QD: Period 1: One 15 mg upadacitinib oral tablet QD for 24 weeks.
- Period 1, 30 mg Cohort: Upadacitinib 30 mg QD: Period 1: One upadacitinib 30 mg oral tablet QD for 24 weeks.
- Period 2, Primary Cohort: Abatacept/Upadacitinib 15 mg QD: Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20. Period 2: open label upadacitinib 15 mg QD for 192 weeks.
- Period 2, Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD: Period 1: One 15 mg upadacitinib oral tablet QD for 24 weeks. Period 2: open label upadacitinib 15 mg QD for 192 weeks.
- Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD: Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20. Period 2: open label upadacitinib 30 mg QD for 192 weeks.
- Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD: Period 1: One upadacitinib 30 mg oral tablet QD for 24 weeks. Period 2: open label upadacitinib 30 mg QD for 192 weeks.
- Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD: Period 1: 500 mg (for body weight <60 kg); 750 mg (for body weight 60-100 kg); and 1000 mg (for body weight >100 kg) IV infusion at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20. Period 2: open label upadacitinib 30 mg QD followed by upadacitinib 15 mg QD for a total of 192 weeks.
- Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD: Period 1: One upadacitinib 30 mg oral tablet QD for 24 weeks. Period 2: open label upadacitinib 30 mg QD followed by upadacitinib 15 mg QD for a total of 192 weeks.
Arm/Group | Period 1, Primary and 30 mg Cohorts: Abatacept | Period 1, Primary Cohort: Upadacitinib 15 mg QD | Period 1, 30 mg Cohort: Upadacitinib 30 mg QD | Period 2, Primary Cohort: Abatacept/Upadacitinib 15 mg QD | Period 2, Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD
All-Cause Mortality (participants affected / at risk) | 1/332 | 2/303 | 0/21 | 7/276 | 16/271 | 0/19 | 0/17 | 1/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 7/332 | 12/303 | 4/21 | 68/276 | 64/271 | 4/19 | 6/17 | 3/12 | 2/12
Other Adverse Events (participants affected / at risk) | 149/332 | 174/303 | 13/21 | 221/276 | 221/271 | 17/19 | 15/17 | 9/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1, Primary and 30 mg Cohorts: Abatacept (N=332) | Period 1, Primary Cohort: Upadacitinib 15 mg QD (N=303) | Period 1, 30 mg Cohort: Upadacitinib 30 mg QD (N=21) | Period 2, Primary Cohort: Abatacept/Upadacitinib 15 mg QD (N=276) | Period 2, Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD (N=271) | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD (N=19) | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD (N=17) | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD (N=12) | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOLVULUS OF SMALL BOWEL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAT NECROSIS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS SOFT TISSUE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BONE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEDICAL DEVICE SITE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CENTRAL OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FRACTURE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-SECRETORY ADENOMA OF PITUITARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN EPITHELIAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCCIPITAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE PHYSICAL PROPERTY ISSUE (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ADNEXA UTERI CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC ORGAN PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRODESIS (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND DRAINAGE (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1, Primary and 30 mg Cohorts: Abatacept (N=332) | Period 1, Primary Cohort: Upadacitinib 15 mg QD (N=303) | Period 1, 30 mg Cohort: Upadacitinib 30 mg QD (N=21) | Period 2, Primary Cohort: Abatacept/Upadacitinib 15 mg QD (N=276) | Period 2, Primary Cohort: Upadacitinib 15 mg QD/Upadacitinib 15 mg QD (N=271) | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD (N=19) | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD (N=17) | Period 2, 30 mg Cohort: Abatacept/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD (N=12) | Period 2, 30 mg Cohort: Upadacitinib 30 mg QD/Upadacitinib 30 mg QD/Upadacitinib 15 mg QD (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (1) | 15 (15) | 10 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 0 (0) | 14 (26) | 9 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TYPE V HYPERLIPIDAEMIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
EYE HAEMATOMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 3 (4) | 0 (0) | 3 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 13 (13) | 8 (9) | 1 (2) | 14 (17) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DUODENOGASTRIC REFLUX (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1) | 11 (14) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 8 (13) | 11 (11) | 2 (2) | 8 (8) | 15 (16) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATIC CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 4 (5) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 3 (3) | 0 (0) | 7 (8) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEELING HOT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 2 (2) | 2 (2) | 6 (9) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 4 (4) | 0 (0) | 11 (11) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ASYMPTOMATIC COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 13 (13) | 8 (8) | 1 (1) | 26 (33) | 16 (18) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 47 (53) | 64 (69) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 3 (3) | 4 (5) | 0 (0) | 10 (16) | 9 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 4 (4) | 12 (14) | 0 (0) | 12 (13) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 35 (35) | 24 (27) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 4 (5) | 0 (0) | 10 (14) | 12 (12) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
LATENT TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 14 (15) | 22 (22) | 1 (1) | 28 (39) | 37 (57) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 4 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIODONTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 8 (9) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 10 (11) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 5 (5) | 5 (6) | 2 (2) | 10 (10) | 7 (9) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 6 (6) | 4 (4) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 (18) | 26 (31) | 0 (0) | 32 (49) | 30 (46) | 5 (5) | 4 (4) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 22 (28) | 20 (27) | 1 (1) | 40 (75) | 40 (67) | 3 (8) | 2 (3) | 1 (1) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BONE CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 14 (15) | 12 (13) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 14 (20) | 0 (0) | 13 (24) | 15 (20) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 12 (18) | 0 (0) | 13 (22) | 17 (28) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 6 (7) | 9 (10) | 0 (0) | 31 (48) | 16 (25) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SCAN ADRENAL GLAND ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 3 (3) | 6 (7) | 0 (0) | 14 (19) | 13 (18) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 5 (6) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 8 (8) | 13 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 8 (8) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 2 (2) | 15 (15) | 15 (16) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6) | 0 (0) | 20 (25) | 18 (20) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GREATER TROCHANTERIC PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 18 (21) | 11 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 15 (15) | 11 (13) | 3 (4) | 32 (57) | 27 (43) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMANGIOMA OF SPLEEN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 10 (11) | 10 (10) | 0 (0) | 12 (17) | 11 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 8 (10) | 6 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AFFECT LABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 10 (14) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER HYPERTROPHY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 2 (2) | 12 (13) | 17 (20) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHOTODERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 11 (11) | 16 (16) | 0 (0) | 25 (27) | 24 (26) | 0 (0) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03086343/Prot_004.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03086343/SAP_005.pdf